CLINICAL TRIAL: NCT03922789
Title: Minimal Important Difference of Walking Test in Subjects With Bronchial Asthma
Status: Completed | Type: Observational
Sponsor: Maugeri Foundation (Other)
Collaborators: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, elisabetta zampogna, Principal Investigator, Maugeri Foundation
Other Study IDs: 2279 CE
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Outcome; Asthma; Pulmonary Rehabilitation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 6 minute walking test — change of 6MWT pre to post pulmonary rehabilitation

SUMMARY:
The Six Minute Walking Test (6MWT) efficiently represents the exercise capacity in subjects with chronic respiratory disease, as asthma. The variation of the walking distance is a parameter used to evaluate the effectiveness of pharmacologic ando non-pharmacologic interventions, as Pulmonary Rehabilitation (PR). However, statistically significant changes in the walking distance do not always represent clinically significant variations.The aim of this prospective study is to determine the Minimal Important Difference (MID) for the 6MWT in subjects affected by asthma, regardless of the severity of the disease.

DETAILED DESCRIPTION:
The Six Minute Walking Test (6MWT) efficiently represents the exercise capacity in subjects with chronic respiratory disease, as asthma. The variation of the walking distance is a parameter used to evaluate the effectiveness of pharmacologic and non-pharmacologic interventions, asPulmonary Rehabilitation (PR). However, statistically significant changes in the walking distance do not always represent clinically significant variations. For this reason, it is important to understand in terms of clinical impact, how to interpret the 6MWT when the walking distance changes over time in the same subject (for example, at the beginning and after PR) or when it differs between subjects (some subjects may improve more and some subjects less). It is not enough to state that the intervention works, it is necessary to say how much it works. The demonstration of a clinically relevant effect must be the primary goal of every treatment. A clinically relevant effect is defined as the minimum achievable benefit, which may lead the medical doctor to change his strategy towards the patient, for example by recommending a particular therapy or treatment. The international scientific community calls the minimum achievable benefit with different names; one of the most common is the Minimal Important Difference (MID). The identification of MID is relevant for the clinician, for the agency that is paying the treatment, for the Regulatory Agency and is equally important for the patient for whose health these groups are responsible. MID for 6MWT has been estimated in subjects with different respiratory diseases and not. In Chronic Obstructive Pulmonary Diseases, a variation of 25 meters is considered significant. Recent studies have shown that asthmatic subjects cover a distance of about 500 meters during 6MWT, and that this distance improves after PR on average of 30-60 meters. Up to-day, however, the 6MWT MID in asthmatic patients has not been investigated.

The aim of this prospective study is to determine the MID for the 6MWT in subjects affected by asthma, regardless of the severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of asthma according to the current guidelines "Global Initiative for Asthma (GINA)
* In therapy with inhaled and/or oral drugs ≥30 days
* Signature of Informed Consent.

Exclusion Criteria:

* Concomitant pathologies with severe short term prognosis.
* Documented Chronic Obstructive Pulmonary Disease diagnosis.
* Inability to perform the 6 Minute Walking Test

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects hospitalized in a Rehabilitation Center to complete a pulmonary rehabilitation programme
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
meters | 20 days
  define the MID for the 6MWT in subjects affected by bronchial asthma of different degrees of severity

SECONDARY OUTCOMES:
Asthma Control Questionnaire (ACQ) | 20 days
  to measure the degree of asthma control. Scores range between 0 (totally controlled) and 6 (severely uncontrolled).
St George Respiratory Questionnaire (SGRQ) | 20 days
  to evaluate the quality of life. Score range 0 (better), 100 (worse)
Chronic Obstructive Pulmonary Disease Assessment Test (CAT) | 20 days
  to evaluate the health status. Score range 0 (better), 40 (worse)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Spanevello, Prof, Study Director — Maugeri Foundation
Locations (1):
- Istituti Clinici Scientifici Maugeri, Tradate, VA, Italy

IPD SHARING:
Plan to Share IPD: Undecided
no decision till now about plan to share